CLINICAL TRIAL: NCT00637078
Title: Evaluation of a Primary Treatment Algorithm Using Combination Therapy for the Management of Patients With Hypertension and Hypercholesterolemia
Brief Title: STITCH2 (Simplified Therapeutic Intervention to Control Hypertension and Hypercholesterolemia)
Acronym: STITCH2
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Western Ontario, Canada (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RPO702
Record Dates: First submitted 2008-03-03; First posted 2008-03-17 (Estimated); Last update posted 2012-06-14 (Estimated); Status verified 2012-06

CONDITIONS: Hypertension; Hypercholesterolemia
Keywords: hypertension; hypercholesterolemia; family physicians; fixed dose combination therapy; cluster randomized controlled trial
MeSH Terms: conditions — Hypertension; Hypercholesterolemia | interventions — Amlodipine; Spironolactone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Drug: Fix dose combination therapy
  Interventions: Other: Treatment algorithm:caduet, Amlodipine, ACEI-ARB combo dose, a-blocker, b-blocker or spironolactone, dyslipidemic therapy with ezetamide
- 2 (No Intervention): Guidelines based management

INTERVENTIONS:
Other: Treatment algorithm:caduet, Amlodipine, ACEI-ARB combo dose, a-blocker, b-blocker or spironolactone, dyslipidemic therapy with ezetamide — initial treatment with a low dose diuretic/ACE-inhibitor or ARB combination followed by a low dose DHP-CCB/statin combination
  Arms: 1

SUMMARY:
The objective of this study is to assess if the implementation of a treatment algorithm including initial treatment with a low dose diuretic/ACE-inhibitor or ARB combination and subsequently a low dose DHP-CCB/statin combination will improve the management of hypertension/hypercholesterolemia compared to guidelines-base management at family practices.

DETAILED DESCRIPTION:
Utilization of fixed dose combination therapy has been advocated as an adherence-enhancing strategy and has been so recommended in the 2007 Canadian Hypertension Education Program (CHEP) recommendations. Further, in a previous study (STITCH) it was demonstrated that a simplified treatment algorithm utilizing initial therapy with a low dose fixed-dose combination therapy improved blood pressure control in hypertensive patients. However, the effectiveness of either a simplified treatment algorithm or the initial use of fixed dose combination therapies for 2 risk factors in hypertensive dyslipidemic patients has yet to be determined. Therefore, the current study is designed to determine whether utilization of a fixed dose combination hypertension/hypercholesterolemia therapy results in improved adherence, patient satisfaction as well as improved rates of reaching target LDL cholesterol and blood pressure.

ELIGIBILITY:
Inclusion Criteria:

* male or female subjects 18 years or older
* documented diagnoses of hypertension and of hypercholesterolemia or current therapy for these conditions
* uncontrolled hypertension (SBP >140 mmHg or DBP >90 mmHg) or cholesterol levels above their threshold based on their global atherosclerotic risk profile (based on ATP III assessment)
* ability to give written informed consent

Exclusion Criteria:

* ischemic heart disease, atrial fibrillation, chronic kidney disease and significant liver disease
* currently prescribed 3 or more drugs to control blood pressure
* currently prescribed 2 or more drugs to control hypercholesterolemia
* participating in other hypertension/hypercholesterolemia studies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Actual)
Dates: Start 2008-02; Primary Completion 2010-06 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects whose systolic BP [SBP] <140 mmHg and diastolic BP [DBP] <90 mmHg)or proportion whose cholesterol levels are at or below threshold based on their global artherosclerotic risk profile compared at the practice level. | 6 months

SECONDARY OUTCOMES:
Secondary measures include the change at 6 months in SBP and DBP and cholesterol levels. These outcomes will be compared at the practice level | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Ross Feldman, MD, Principal Investigator — Deputy Director; George Dresser, MD, Principal Investigator — Co prinicipal investigator
Locations (1):
- Robarts Research Insititute, London, Ontario, Canada